CLINICAL TRIAL: NCT03218176
Title: Tourniquets Type Combat Application Tourniquet (CAT): Vascular Suffering According to the Proximal or Distal Location, Simple or Staggered. Study to Upper and Lower Limbs
Brief Title: Tourniquets Type Combat Application Tourniquet: Proximal or Distal Location, Simple or Staggered on Upper and Lower Limb
Acronym: GARROTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: GARROTS (29BRC17.0087)
Record Dates: First submitted 2017-07-10; First posted 2017-07-14 (Actual); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Hemorrhage
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Proximal single upper limb (Active Comparator): Laying a single tourniquet on the root of the upper limb
  Interventions: Device: Proximal single upper limb
- Proximal staggered upper limb (Experimental): Laying two staggered tourniquets : one on the root of the upper limb and a second 5 cm below the previous one
  Interventions: Device: Proximal staggered upper limb
- Distal single upper limb (Experimental): Laying a single tourniquet on the forearm
  Interventions: Device: Distal single upper limb
- Distal staggered upper limb (Experimental): Laying two staggered tourniquets : one on the forearm and a second 5 cm below the previous one
  Interventions: Device: Distal staggered upper limb
- Proximal single lower limb (Active Comparator): Laying a single tourniquet on the root of the lower limb
  Interventions: Device: Proximal single lower limb
- Proximal staggered lower limb (Experimental): Laying two staggered tourniquets : one on the root of the lower limb and a second 5 cm below the previous one
  Interventions: Device: Proximal staggered lower limb
- Distal single lower limb (Experimental): Laying a single tourniquet on the calf
  Interventions: Device: Distal single lower limb
- Distal staggered lower limb (Experimental): Laying two staggered tourniquets : one on the calf and a second 5 cm below the previous one
  Interventions: Device: Distal staggered lower limb

INTERVENTIONS:
Device: Proximal single upper limb — Measurement of pain, pressure under tourniquet, feeling and abolition of pulse doppler and pulse oximetry
  Arms: Proximal single upper limb
Device: Proximal staggered upper limb — Measurement of pain, pressure under tourniquet, feeling and abolition of pulse doppler and pulse oximetry
  Arms: Proximal staggered upper limb
Device: Distal single upper limb — Measurement of pain, pressure under tourniquet, feeling and abolition of pulse doppler and pulse oximetry
  Arms: Distal single upper limb
Device: Distal staggered upper limb — Measurement of pain, pressure under tourniquet, feeling and abolition of pulse doppler and pulse oximetry
  Arms: Distal staggered upper limb
Device: Proximal single lower limb — Measurement of pain, pressure under tourniquet, feeling and abolition of pulse doppler and pulse oximetry
  Arms: Proximal single lower limb
Device: Proximal staggered lower limb — Measurement of pain, pressure under tourniquet, feeling and abolition of pulse doppler and pulse oximetry
  Arms: Proximal staggered lower limb
Device: Distal single lower limb — Measurement of pain, pressure under tourniquet, feeling and abolition of pulse doppler and pulse oximetry
  Arms: Distal single lower limb
Device: Distal staggered lower limb — Measurement of pain, pressure under tourniquet, feeling and abolition of pulse doppler and pulse oximetry
  Arms: Distal staggered lower limb

SUMMARY:
A tourniquet is used to stop abundant bleeding when simple compression is not effective. The investigators will study the vascular suffering of the tourniquets according to their location on the limb: limb (arm / thigh) or distal (forearm / leg). Vascular suffering will be evaluated by the loss of the radial doppler flux for the tourniquets placed on the upper limb and in the tibial anterior to the lower limb by the loss of the pulse oximetry pulse and the collection of the signs described by the volunteers (pain, Paresthesia, cold sensation).

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years (major)
* Volunteer to participate in research

Exclusion Criteria:

* Age less than 18 years
* Known coagulation disorder
* Known vascular disorder
* Known neurological disorder of the limbs
* Known muscle disorders of the limbs
* Presence of an implant in one of the limbs (vascular, contraceptive ...)
* Simultaneous participation in research involving anticoagulant therapy
* History of phlebitis
* Persons of full age who are subject to legal protection (safeguard of justice, person placed in curatorship, guardianship), persons deprived of their liberty.
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2017-10-23 (Actual); Study Completion 2017-10-23 (Actual)

PRIMARY OUTCOMES:
Upper limb : Assessment of Pain by Digital Evaluation (EN) after 10 min of compression | 10 min
  The main evaluation criterion for the superior member is the assessment of the pain felt according to the location of the tourniquets at the time of laying and at 10min. For the same location of tourniquet, the pain caused by the laying of one versus two tourniquets will be compared. For proximal versus distal, comparisons will be made for 1 tourniquet and for staggered tourniquets.
Lower limb : Pressure (mmHg) needed to abolish the pulse | 10 min
  The main evaluation criterion for the inferior member is the pressure under the tourniquet, necessary to obtain an abolition of the anterior tibial pulse (measured in Doppler). By means of a balloon connected to a pressure gauge and fixed under each tourniquet, a measure of the pressure exerted (in mmHg) by the tourniquet (s) on the skin will be measured at laying. The comparison will be made for each type of pose (single vs stage) between the proximal and distal layers.

SECONDARY OUTCOMES:
Lower limb pain | 10 min
  The pain will be relieved according to the Digital Scale at the time of the raising of the tourniquets and at 10 minutes. For the same location of tourniquet, the pain caused by the laying of one versus two tourniquets will be compared. For proximal versus distal, comparisons will be made for 1 tourniquet and for staggered tourniquets.
Upper limb pressure under tourniquet | 10 min
  By means of a balloon connected to a pressure gauge and fixed under each tourniquet, a measure of the pressure exerted (in mmHg) by the tourniquet (s) on the skin will be measured at laying. The comparison will be made for each type of pose (single vs staggered) between the proximal and distal layers.
Pulse oximetry | 10 min
  Evaluation of the loss of the pulse oximetry, by a pulse oximeter placed on the finger or the toe, according to each mode of pose
Loss of arterial Doppler pulse | 10 min
  The loss of the Doppler signal on the radial artery for the upper limbs and on the tibial anterior artery for the lower limbs will be evaluated for each type of poses to confirm arterial occlusion for each type of pose.

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Gelin, MD, Principal Investigator — CHU de Brest
Locations (1):
- CHU de Brest, Brest, France